CLINICAL TRIAL: NCT04216017
Title: A Randomized Controlled Pilot Study Evaluating the Efficacy of Early Glenohumeral Cortisone Injection in Patients With Shoulder Stiffness Following Proximal Humerus Fractures
Brief Title: Glenohumeral Cortisone Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Jonah Hebert-Davies, Assistant Professor, School of Medicine: Orthopedics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00007576; P30AR072572 (NIH)
Record Dates: First submitted 2019-12-24; First posted 2020-01-02 (Actual); Results first posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-08

CONDITIONS: Humeral Fractures
MeSH Terms: conditions — Humeral Fractures | interventions — Triamcinolone Acetonide; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Controls (Placebo Comparator): Patients receiving lidocaine
  Interventions: Drug: Lidocaine
- Cases (Active Comparator): Patients receiving Kenalog
  Interventions: Drug: kenalog

INTERVENTIONS:
Drug: kenalog — Cortisone injection into shoulder
  Arms: Cases
Drug: Lidocaine — Lidocaine injection into shoulder
  Arms: Controls

SUMMARY:
The objective of this project is to determine if giving a cortisone injection to patients with proximal humerus fractures who have stiff shoulders recover their range of motion.

DETAILED DESCRIPTION:
THis is a randomized control trial to determine if giving a cortisone injection to patients with proximal humerus fractures who have stiff shoulders recover their range of motion.

ELIGIBILITY:
Inclusion Criteria:

1.18-90

2. Proximal Humerus Fracture

3. Decreased range of motion at 6 wk follow-up

4. Likely to be available for follow up for 26 wks

Exclusion Criteria:

1. Known drug allergy to kenalog or lidocaine
2. Unable to complete functional outcome
3. Pregnant Women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonah Hebert-Davies, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Controls | Cases
Started | 5 | 4
Completed | 4 | 4
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Controls | Cases | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9
ASES [Mean (Standard Deviation); unit: units on a scale] — American Shoulder Elbow Society Score The ASES is a condition-specific scale that is intended to measure functional limitations and pain of the shoulder.0 (worst-100 (best)
  units on a scale | 43.4 (19.3) | 51.3 (5.4) | 46.9 (14.9)

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder Elbow Society Score
Description: Outcome Instrument high is good low is bad 0-100 The ASES is a condition-specific scale that is intended to measure functional limitations and pain of the shoulder.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Controls | Cases
Number analyzed (Participants) | 4 | 4
score on a scale | 46 (20) | 87 (8)

2. Secondary Outcome: Visual Analogue Scale
Description: pain scale - high is bad - low is good 0-100
Time Frame: 24 weeks
Population: Population at 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controls | Cases
Number analyzed (Participants) | 4 | 4
units on a scale | 4 (3.7) | 1 (0.8)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Controls | Cases
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT04216017/Prot_002.pdf
  • Informed Consent Form (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT04216017/ICF_001.pdf